CLINICAL TRIAL: NCT04022941
Title: Efficacy and Safety of Sodium Benzoate in the Management of Hyperammonemia in Infants, Children and Adolescents With Chronic Liver Disese - A Randomised Controlled Trial.
Brief Title: Efficacy and Safety of Sodium Benzoate in the Management of Hyperammonemia in Infants, Children and Adolescent With Chronic Liver Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-22
Record Dates: First submitted 2019-07-07; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Chronic Liver Disease
MeSH Terms: interventions — Sodium Benzoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Benzoate (Experimental): Group A will receive drug packets containing 2.5 gm sodium benzoate and 5 gm powdered table sugar for 5days.
  Interventions: Drug: Sodium Benzoate
- Placebo (Placebo Comparator): Group B will receive 7.5 gm packets of powdered table sugar for 5 days as placebo which is similar in appearance and taste as sodium benzoate.
  Interventions: Other: Powdered table sugar as palcebo

INTERVENTIONS:
Drug: Sodium Benzoate — Group A will receive drug packets containing 2.5 gm sodium benzoate and 5 gm powdered table sugar for 5 days.
  Arms: Sodium Benzoate
Other: Powdered table sugar as palcebo — Group B will receive 7.5 gm packets of powdered table sugar for 5 days as placebo which is similar in appearance and taste as sodium benzoate.
  Arms: Placebo

SUMMARY:
Subject will be randomize in two groups. Group A will receive drug packets containing 2.5 gm sodium benzoate and 5 gm powdered table sugar for 5days.Since the dosage of Sodium Benzoate is Sta t250mg/Kg and then 250mg/Kg in next 24 hours, each patient would be given 750mg /kg stat and 750mg /kg in next 24 hours,keeping in view that 2/3 of powder used would be powdered sugar in the intervention arm. The dose of the powder used would be doubled in case of the ammonia level more than 300 mcg/dl. The drug will be prepared in sterile water and administered per orally or via the nasogastric tube. All the enrolled patients would be treated with SMT as per the recommendations of the EASL/AASLD 2014 guidelines of management of hepatic encephalopathy.

Group B will receive 7.5 gm packets of powdered table sugar for 5 days as placebo which is similar in appearance and taste as sodium benzoate.

ELIGIBILITY:
Inclusion Criteria:

- Infants, children and adolescents under 18 years of age with decompensated Chronic liver disease with hyperammonemia < 400 mcgm and /dl.

Exclusion Criteria:

1. Patients who have received sodium benzoate within 1 week priorto evaluation.
2. Baseline serum sodium above 155 mEq/L
3. Patients with Grade 3 ascites as per IAC classification.
4. Patients who did not give a written informed consent.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the blood ammonia levels at 5 days of starting therapy in both groups. | Day 5

SECONDARY OUTCOMES:
Change in the grading of Hepatic Encephalopathy in both groups. | Day 28
Change in the grading of Hepatic Encephalopathy in both groups. | Day 90
Proportion of children with worsening ascites in both groups. | Day 28
Proportion of children with worsening ascites in both groups. | Day 90
Proportion of children with hypernatremia in both groups. | Day 28
Proportion of children with hypernatremia in both groups. | Day 90
Proportion of children with metabolic acidosis in both groups. | Day 28
Proportion of children with metabolic acidosis in both groups. | Day 90
Duration of hospital stay in both groups. | Day 28
Duration of hospital stay in both groups. | Day 90
Short term survival with native liver in both groups | Day 28
Short term survival with native liver in both groups | Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India